CLINICAL TRIAL: NCT02726724
Title: Does the Presence of Observers Influence the Success of the Neonatal Endotracheal Intubation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Dr Brahim Bensouda, MD, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Hopital Maisonneuve Rosemont
Record Dates: First submitted 2016-03-22; First posted 2016-04-04 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Stress
Keywords: Stress-Resident performance-Observers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Condition B (Experimental): An audience of 5 people with at least 2 neonatologists will be present with the operator during the intubation of the mannequin.
  Interventions: Other: 5 observers
- Condition A (Experimental): Only the staff will be present with the operator during the intubation of the mannequin.
  Interventions: Other: 1 observer

INTERVENTIONS:
Other: 5 observers
  Arms: Condition B
Other: 1 observer
  Arms: Condition A

SUMMARY:
The Endotracheal intubation (ETI) of a neonate is a procedure that usually attracts a large number of observers. The fear of being judged by others could cause an increased level of stress, especially on the junior trainees. Little research has focused on the effect of the audience on the level of stress and therefore, on the success rate of complicated procedures in neonatal intensive care.

Hypothesis:Investigators hypothesize that time to successful intubation (in seconds) will be longer with the presence of observers.

DETAILED DESCRIPTION:
Objective: The aim of this study will be to provide objective evidence supporting that junior trainees are less successful at neonatal ETI when in the presence of a large audience. If this hypothesis is correct, this data will provide evidence to support the residents request for less people around during the procedure, which may increase the chance of a successful intubation.

After Investigators obtained written consent - the selected student-will be asked to wear a cardiac monitor and 5 minutes later after a period of rest, they will be called in the delivery room. Two minutes after their arrival they will be given a stylet and a 3.5 ET tube and will be asked to intubate orally a mannequin, after 30 seconds, the operator will be reminded of the time. After 45 seconds the attempts will be stopped.

Participants will be informed of their right to discontinue participation at any time. The trainee will be informed at the end of the experience about the aim of the study and will be asked to keep it confidential.

The trainees will be randomized in two groups that differentiate in the conditions under which they will start the intubation.

Condition A: Only the staff will be present with the operator Condition B: An audience of 5 people with at least 2 neonatologists will be present in case of junior resident or the responsible of stage in case of respiratory therapy students.

The residents who performed intubation in condition A will do a repeat intubation 24 hours later using condition B and vice versa. The time and the local of the 2 procedures will be the same in both conditions.

Time to successful intubation will be compared between the two experimental conditions for each subject with paired t test. A p<0.05 will be considered significant.

To estimate the required sample size, Investigators used the study O'Donnel and al who gave an approximate intubation time for trainees of 38 seconds with standard deviation of 20 seconds (14). Using an alpha threshold of 0.05 and power of 80 %, a sample size of 51 subjects is required to detect 8 second difference time between the two different groups. Eight seconds represents a 25 % change in time to intubate and is clinically significant for a newborn.

ELIGIBILITY:
Inclusion Criteria:

* Junior residents during the first year of residency and respiratory therapy students who never had any experience with a real newborn intubation will participate to the studies. The mannequin used during the procedure is the same for all the students and is different from what they used during there training before starting the rotation in the NICU.

Exclusion Criteria:

* Students with a history of beta blockers within in the past year and students with a history of antidepressant medication are excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Evaluating the differences in the duration (seconds) to reach intubation of the mannequin between the two experimental conditions. | 24 hour
  The duration of each individual attempt will be recorded as the time in seconds from insertion of the laryngoscope into the mouth to its removal.

SECONDARY OUTCOMES:
Variability of the heart rate of the operator between the condition A and B. | 24 hour
  After investigators obtained written consent - the selected student-will be asked to wear a cardiac monitor. The heart rate will be recorded before, during and after the end of the mannequin intubation. The variability in percentage during the intubation between the condition A and B will be compared.
The number of wrong ET length position between the condition A and B | 24 hour
  Length of the position of the tube will be assessed 10 seconds after the intubation. Any position above 10 cm and bellow 8 cm will be considered wrong. The number of wrong ET length position between the condition A and B will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Brahim BB Bensouda, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hopital Maisonneuve Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bensouda B, Mandel R, Mejri A, Lachapelle J, St-Hilaire M, Ali N. Effect of an audience on trainee stress and performance during simulated neonatal intubation: a randomized crossover trial. BMC Med Educ. 2018 Oct 3;18(1):230. doi: 10.1186/s12909-018-1338-4. PMID 30285715